CLINICAL TRIAL: NCT00440466
Title: A Randomized, Open-label, Multicenter Study of Epoetin Alfa Comparing Two Extended Dosing Regimens, Once-every-two-weeks and Once-every-four-weeks, With the Once-weekly Dosing Regimen for Maintenance Treatment in Anemic Subjects With Chronic Kidney Disease
Brief Title: PROCRIT Extended Dosing For Maintenance of Hemoglobin in Pre-Dialysis CKD Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR010414; EPOAKD3002
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Results first posted 2011-04-14 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Anemia; Renal Diseases
Keywords: Anemia; Reduction in the number of erythrocytes; Hemoglobin low level; Red blood cell deficiency; Procrit; Epoetin alfa; Chronic kidney disease
MeSH Terms: conditions — Anemia; Kidney Diseases; Renal Insufficiency, Chronic | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 001 (Experimental): epoetin alfa Continue pre-study once weekly dose of epoetin alfa for 36 weeks
  Interventions: Drug: epoetin alfa
- 003 (Experimental): epoetin alfa Quadruple the pre-study once weekly dose of epoetin alfa every 4 weeks for 36 wk
  Interventions: Drug: epoetin alfa
- 002 (Experimental): epoetin alfa Double the pre-study once weekly dose of epoetin alfa every 2 weeks for 36 wks
  Interventions: Drug: epoetin alfa

INTERVENTIONS:
Drug: epoetin alfa — Continue pre-study once weekly dose of epoetin alfa for 36 weeks
  Arms: 001
Drug: epoetin alfa — Double the pre-study once weekly dose of epoetin alfa every 2 weeks for 36 wks
  Arms: 002
Drug: epoetin alfa — Quadruple the pre-study once weekly dose of epoetin alfa every 4 weeks for 36 wk
  Arms: 003

SUMMARY:
The purpose of this study is to demonstrate that once every-2-weeks and once every-4-weeks treatment with epoetin alfa, a drug that increases red blood cell production, in patients with anemia associated with chronic kidney disease, is not less effective than treatment with epoetin alfa that is given once a week

DETAILED DESCRIPTION:
A consequence of chronic kidney disease is anemia due to decreased production of erythropoietin. Anemia is associated with decreased oxygen delivery and utilization, and can result in fatigue, lethargy, decreased cognition and mental acuity, and cardiac complications.This study was designed to compare 2 dosing regimens, once every-2-weeks and once every-4-weeks with the once-weekly dosing regimen. Men and women who are diagnosed with anemia associated with chronic kidney disease will participate in this study. Approximately 400 patients will be included. This is a randomized (patients are assigned different treatments based on chance), open-label, multicenter study of epoetin alfa in patients who are not on dialysis and who are already maintaining anemia with epoetin alfa administered once weekly. The study is 40 to 42 weeks in duration. All eligible patients will be treated with epoetin alfa according to one of the following 3 regimens: once-a-week injection (Group 1), or once every-2-weeks injection (Group 2), or once every-4-weeks injection (Group 3). The maximum volume per injection will not be more than 1 mL, therefore some patients may receive more than one injection per dose. The study treatment includes a period to convert to the new dosing regimen, and a subsequent stable maintenance treatment period. After the initial dose, hemoglobin will be measured on a weekly basis and used to determine adjustments in dose for each patient. The primary hypothesis is that the average change in hemoglobin level in the groups that received epoetin alfa once every 2 weeks or once every 4 weeks is not lower than the change in hemoglobin level in the group that received epoetin alfa only once a week. Adverse events will be monitored throughout the study. Clinical laboratory examinations, vital signs, and physical examinations will be conducted routinely to ensure patient safety. Approximately 1 mL of epoetin alfa will be injected under the skin either once a week, once every 2 weeks, or once every 4 weeks (maximum doses of 20,000 IU once a week, 40, 000 IU every 2 weeks, or 80,000 IU every 4 weeks, respectively) for up to 36 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for chronic kidney disease, defined as a glomerular filtration rate (GFR) >=15 mL/min per 1.73 m2 and <60 mL/min per 1.73 m2 (Stages 3 and 4) as calculated by the central laboratory
* Hemoglobin level between 10.0 and 11.9 g/dL during the 4 weeks before randomization
* History of increase in hemoglobin after the initial dose
* Stable dose of epoetin alfa given once-weekly before randomization.

Exclusion Criteria:

* Uncontrolled hypertension
* Iron deficiency
* iron overload
* severe congestive heart failure
* Active infection
* Recent heart attack, Stroke or blood clot.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2007-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (66):
- United States (66):
  - Chula Vista, California
  - Fountain Valley, California
  - Los Angeles, California
  - Lynwood, California
  - Orange, California
  - Riverside, California
  - San Dimas, California
  - West Hills, California
  - Yuba City, California
  - Lakewood, Colorado
  - Thornton, Colorado
  - Washington D.C., District of Columbia
  - Clearwater, Florida
  - Miami, Florida
  - Pembroke Pines, Florida
  - Plantation, Florida
  - Springhill, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Zephyrhills, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Macon, Georgia
  - Chicago, Illinois
  - Evergreen Park, Illinois
  - Peoria, Illinois
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Methuen, Massachusetts
  - Plymouth, Massachusetts
  - Springfield, Massachusetts
  - Detroit, Michigan
  - Flint, Michigan
  - Picayune, Mississippi
  - St Louis, Missouri
  - Great Neck, New York
  - New York, New York
  - Springfield Gardens, New York
  - Charlotte, North Carolina
  - Greenville, North Carolina
  - Monroe, North Carolina
  - Dayton, Ohio
  - Maumee, Ohio
  - Allentown, Pennsylvania
  - Doylestown, Pennsylvania
  - Erie, Pennsylvania
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Wynnewood, Pennsylvania
  - Providence, Rhode Island
  - Bamberg, South Carolina
  - Columbia, South Carolina
  - Orangeburg, South Carolina
  - Rock Hill, South Carolina
  - Sumter, South Carolina
  - Arlington, Texas
  - Fountain Valley, Texas
  - Houston, Texas
  - Longview, Texas
  - San Antonio, Texas
  - Fairfax, Virginia
  - Hampton, Virginia
  - Petersburg, Virginia
  - Richmond, Virginia
  - Tacoma, Washington

REFERENCES:
- See also: A Randomized, Open-label, Multicenter Study of Epoetin Alfa Comparing Two Dosing Regimens, Once-every-two-weeks and Once-every-four-weeks, with Once-weekly Dosing Regimen for Maintenance Treatment in Anemic Subjects with Chronic Kidney Disease — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=58&filename=CR010414_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Epoetin Alfa QW: Continue pre-study once weekly dose of epoetin alfa for 36 weeks
- Epoetin Alfa Q2W: Double the pre-study once weekly dose of epoetin alfa every 2 weeks for 36 wks
- Epoetin Alfa Q4W: Quadruple the pre-study once weekly dose of epoetin alfa every 4 weeks for 36 wk
Period: Overall Study
Arm/Group | Epoetin Alfa QW | Epoetin Alfa Q2W | Epoetin Alfa Q4W
Started | 108 | 107 | 215
Completed | 95 | 92 | 174
Not Completed | 13 | 15 | 41
Not completed — Death | 3 | 2 | 9
Not completed — Adverse Event | 3 | 4 | 11
Not completed — Lost to Follow-up | 1 | 0 | 2
Not completed — Physician Decision | 2 | 0 | 1
Not completed — Protocol Violation | 2 | 0 | 4
Not completed — Withdrawal by Subject | 2 | 5 | 9
Not completed — Began Dialysis | 0 | 0 | 1
Not completed — Met Hemoglobin Withdrawal Criteria | 0 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epoetin Alfa QW | Epoetin Alfa Q2W | Epoetin Alfa Q4W | Total
Number analyzed (Participants) | 108 | 107 | 215 | 430
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 33 | 26 | 57 | 116
  >=65 years | 75 | 81 | 158 | 314
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (13.04) | 71.7 (10.63) | 71.1 (12.48) | 71 (12.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 73 | 126 | 267
  Male | 40 | 34 | 89 | 163

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin Concentration in Grams Per Deciliter (g/dL) From Baseline to the Average of the Last 12 Weeks of Treatment
Time Frame: from baseline (Week 1) to the last 12 weeks of treatment
Population: Modified Intent-To-Treat (mITT) population defined as all participants who were randomly assigned to treatment with epoetin alfa and had at least 1 post-randomization hemoglobin assessment.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Epoetin Alfa QW | Epoetin Alfa Q2W | Epoetin Alfa Q4W
Number analyzed (Participants) | 107 | 105 | 215
g/dL | -0.02 (0.728) | -0.10 (0.774) | -0.19 (0.738)
Statistical Analysis 1: Comparison: Epoetin Alfa QW vs Epoetin Alfa Q2W; The null hypothesis was that the lower limit of the 95% confidence interval (CI) for the difference in mean change in hemoglobin from baseline to the average of the last 12 weeks of treatment between the every-2-weeks (Q2W) and once-weekly (QW) groups would be lower than -1 g/dL; Test type: Non-Inferiority or Equivalence — Assuming a difference in the mean change in hemoglobin from baseline to the average of the last 12 weeks of treatment of -0.3 g/dL between QW and Q2W groups, a pooled standard deviation of 1.5 g/dL, and a noninferiority margin of 1 g/dL, a sample size of approximately 200 subjects (100 per group) would provide 90% power to demonstrate that Q2W group would not inferior to QW group for an overall 2-sided 0.05 significance level; ANCOVA; Difference of Least Squares Means = -0.03, 95% CI 2-sided [-0.208 to 0.153], Standard Error of Mean 0.092
Statistical Analysis 2: Comparison: Epoetin Alfa QW vs Epoetin Alfa Q4W; The null hypothesis was that the lower limit of the 95% confidence interval (CI) for the difference in mean change in hemoglobin from baseline to the average of the last 12 weeks of treatment between the every-4-weeks (Q4W) and once-weekly (QW) groups would be lower than -1 g/dL; Test type: Non-Inferiority or Equivalence — Under the same assumptions in the sample size calculation for the QW and the Q2W, 100 subjects would be needed for the Q4W. However, because Study EPO-AKD-3001 and the current study both included QW and Q2W groups, the sample size would add up to 200 for each group if combined, the sample size in the Q4W group in the current study was increased to 200 subjects in order to enroll a comparable and sufficiently large number of subjects in each of the 3 extended dosing groups across the 2 studies; ANCOVA; Difference of Least Squares Means = -0.09, 95% CI 2-sided [-0.249 to 0.063], Standard Error of Mean 0.079

2. Secondary Outcome: Proportion of Weeks Per Patient With Hemoglobin Concentration Between 10.0 and 11.9 Grams Per Deciliter (g/dL)
Time Frame: Weeks 13-37
Population: as for outcome 1
Measure: Median (Full Range); unit: Proportion
Arm/Group | Epoetin Alfa QW | Epoetin Alfa Q2W | Epoetin Alfa Q4W
Number analyzed (Participants) | 97 | 100 | 200
Proportion | 0.87 [0.3 to 1.0] | 0.88 [0.0 to 1.0] | 0.83 [0.0 to 1.0]

3. Other Pre Specified Outcome: Participants Who Exceeded a Hemoglobin Concentration of 11.9 Grams Per Deciliter (g/dL)
Time Frame: 36 weeks of treatment
Population: Safety population defined as all participants who received at least 1 injection of study drug
Measure: Number; unit: Participants
Arm/Group | Epoetin Alfa QW | Epoetin Alfa Q2W | Epoetin Alfa Q4W
Number analyzed (Participants) | 107 | 105 | 215
Participants | 79 | 89 | 161
Statistical Analysis 1: Comparison: Epoetin Alfa QW vs Epoetin Alfa Q2W; Test type: Superiority or Other; 95% Confidence Interval; Difference in percentage of participants = 10.9, 95% CI 2-sided [0.1 to 21.7]
Statistical Analysis 2: Comparison: Epoetin Alfa QW vs Epoetin Alfa Q4W; Test type: Superiority or Other; 95% of Confidence Interval; Difference in percentage of participants = 1.1, 95% CI 2-sided [-9.1 to 11.2]

4. Other Pre Specified Outcome: Maximum Hemoglobin Concentration in Grams Per Deciliter (g/dL)
Time Frame: 36 weeks of treatment
Population: Safety population defined as all participants who received at least 1 injection of study drug
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Epoetin Alfa QW | Epoetin Alfa Q2W | Epoetin Alfa Q4W
Number analyzed (Participants) | 107 | 105 | 215
g/dL | 12.35 (0.828) | 12.48 (0.760) | 12.46 (0.988)
Statistical Analysis 1: Comparison: Epoetin Alfa QW vs Epoetin Alfa Q2W; Test type: Superiority or Other; ANOVA; Difference in Least Squares Means = 0.13, 95% CI 2-sided [-0.113 to 0.372]
Statistical Analysis 2: Comparison: Epoetin Alfa QW vs Epoetin Alfa Q4W; Test type: Superiority or Other; ANOVA; Difference in Least Squares Means = 0.11, 95% CI 2-sided [-0.098 to 0.320]

5. Other Pre Specified Outcome: Participants Who Met or Exceeded 1.0 Grams Per Deciliter Per 2 Weeks (g/dL/2 Weeks) Hemoglobin Rates of Rise
Time Frame: 36 weeks of treatment
Population: Safety population defined as all participants who received at least 1 injection of study drug
Measure: Number; unit: Particpants
Arm/Group | Epoetin Alfa QW | Epoetin Alfa Q2W | Epoetin Alfa Q4W
Number analyzed (Participants) | 107 | 105 | 215
Particpants | 84 | 91 | 191
Statistical Analysis 1: Comparison: Epoetin Alfa QW vs Epoetin Alfa Q2W; Test type: Superiority or Other; 95% of Confidence Interval; Difference in percentage of participants = 8.2, 95% CI 2-sided [-2.0 to 18.3]
Statistical Analysis 2: Comparison: Epoetin Alfa QW vs Epoetin Alfa Q4W; Test type: Superiority or Other; 95% of Confidence Interval; Difference in percentage of participants = 10.3, 95% CI [1.5 to 19.2]

6. Other Pre Specified Outcome: Participants Who Met or Exceeded 1.5 Grams Per Deciliter Per 2 Weeks (g/dL/2 Weeks) Hemoglobin Rates of Rise
Time Frame: 36 weeks of treatment
Measure: Number; unit: Participants
Arm/Group | Epoetin Alfa QW | Epoetin Alfa Q2W | Epoetin Alfa Q4W
Number analyzed (Participants) | 107 | 105 | 215
Participants | 52 | 57 | 124
Statistical Analysis 1: Comparison: Epoetin Alfa QW vs Epoetin Alfa Q2W; Test type: Superiority or Other; 95% of Confidence Interval; Difference in percentage of participants = 5.7, 95% CI 2-sided [-7.7 to 19.1]
Statistical Analysis 2: Comparison: Epoetin Alfa QW vs Epoetin Alfa Q4W; Test type: Superiority or Other; 95% of Confidence Interval; Difference in percentage of participants = 9.1, 95% CI 2-sided [-2.5 to 20.6]

7. Other Pre Specified Outcome: Participants Who Met or Exceeded 2.0 Grams Per Deciliter Per 2 Weeks (g/dL/2 Weeks) Hemoglobin Rates of Rise
Time Frame: 36 weeks of treatment
Population: Safety population defined as all participants who received at least 1 injection of study drug
Measure: Number; unit: Participants
Arm/Group | Epoetin Alfa QW | Epoetin Alfa Q2W | Epoetin Alfa Q4W
Number analyzed (Participants) | 107 | 105 | 215
Participants | 37 | 33 | 68
Statistical Analysis 1: Comparison: Epoetin Alfa QW vs Epoetin Alfa Q2W; Test type: Superiority or Other; 95% of Confidence Interval; Difference in percentage of participants = -3.2, 95% CI 2-sided [-15.8 to 9.5]
Statistical Analysis 2: Comparison: Epoetin Alfa QW vs Epoetin Alfa Q4W; Test type: Superiority or Other; 95% of Confidence Interval; Difference in percentage of participants = -3.0, 95% CI 2-sided [-13.9 to 8.0]

8. Other Pre Specified Outcome: Maximum Hemoglobin Rate of Rise in Grams Per Deciliter (g/dL/2 Weeks)
Time Frame: 36 weeks of treatment
Population: Safety population defined as all participants who received at least 1 injection of study drug
Measure: Mean (Standard Deviation); unit: g/dL/2 weeks
Arm/Group | Epoetin Alfa QW | Epoetin Alfa Q2W | Epoetin Alfa Q4W
Number analyzed (Participants) | 107 | 105 | 215
g/dL/2 weeks | 1.77 (1.068) | 1.69 (0.790) | 1.81 (1.173)
Statistical Analysis 1: Comparison: Epoetin Alfa QW vs Epoetin Alfa Q2W; Test type: Superiority or Other; ANOVA; Difference in Least Squares Means = -0.08, 95% CI [-0.367 to 0.208]
Statistical Analysis 2: Comparison: Epoetin Alfa QW vs Epoetin Alfa Q4W; Test type: Superiority or Other; ANOVA; Difference in Least Squares Means = 0.04, 95% CI 2-sided [-0.206 to 0.289]

9. Other Pre Specified Outcome: Number of Participants Who Died
Time Frame: 36 weeks of treatment
Measure: Number; unit: Participants
Arm/Group | Epoetin Alfa QW | Epoetin Alfa Q2W | Epoetin Alfa Q4W
Number analyzed (Participants) | 108 | 107 | 215
Participants | 4 | 3 | 9

ADVERSE EVENTS:
Arm/Group | Epoetin Alfa QW | Epoetin Alfa Q2W | Epoetin Alfa Q4W
Serious Adverse Events (participants affected / at risk) | 24/108 | 28/107 | 56/215
Other Adverse Events (participants affected / at risk) | 59/108 | 59/107 | 116/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epoetin Alfa QW (N=108) | Epoetin Alfa Q2W (N=107) | Epoetin Alfa Q4W (N=215)
Anaemia (Blood and lymphatic system disorders) | 2 | 4 | 1
Hypercoagulation (Blood and lymphatic system disorders) | 1 | 0 | 0
Splenic cyst (Blood and lymphatic system disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 5 | 8 | 4
Myocardial infarction (Cardiac disorders) | 2 | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 2
Cardiac failure (Cardiac disorders) | 1 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 2
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 1
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 | 1 | 0
Gastric mucosal lesion (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 4 | 2 | 3
Asthenia (General disorders) | 1 | 0 | 1
Sudden cardiac death (General disorders) | 2 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1
Gallbladder disorder (Hepatobiliary disorders) | 0 | 1 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 3
Pneumonia (Infections and infestations) | 0 | 1 | 2
Bronchitis (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Viral infection (Infections and infestations) | 2 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Intervertebral discitis (Infections and infestations) | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 1
Pharyngeal abscess (Infections and infestations) | 0 | 1 | 0
Sepsis syndrome (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 2
Blood creatinine increased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 3
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 3
Syncope (Nervous system disorders) | 1 | 0 | 2
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 2
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Cervical cord compression (Nervous system disorders) | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Vascular dementia (Nervous system disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 5 | 5 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 2 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 2
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 3
Aortic aneurysm (Vascular disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1
Hypertensive crisis (Vascular disorders) | 1 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 2
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 1
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Epoetin Alfa QW (N=108) | Epoetin Alfa Q2W (N=107) | Epoetin Alfa Q4W (N=215)
Anaemia (Blood and lymphatic system disorders) | 6 | 5 | 10
Diarrhoea (Gastrointestinal disorders) | 8 | 5 | 14
Constipation (Gastrointestinal disorders) | 5 | 5 | 15
Vomiting (Gastrointestinal disorders) | 6 | 6 | 10
Nausea (Gastrointestinal disorders) | 3 | 6 | 12
Oedema (General disorders) | 5 | 13 | 16
Oedema peripheral (General disorders) | 6 | 10 | 14
Fatigue (General disorders) | 6 | 5 | 15
Urinary tract infection (Infections and infestations) | 12 | 8 | 13
Nasopharyngitis (Infections and infestations) | 4 | 6 | 15
Upper respiratory tract infection (Infections and infestations) | 7 | 6 | 9
Hyperkalaemia (Metabolism and nutrition disorders) | 7 | 7 | 18
Gout (Metabolism and nutrition disorders) | 6 | 4 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 5 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 5 | 7
Dizziness (Nervous system disorders) | 3 | 7 | 18
Headache (Nervous system disorders) | 5 | 6 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 15
Hypertension (Vascular disorders) | 11 | 14 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the only disclosure restriction on the PI is that the sponsor has 60 days to review results communications prior to public release and can embargo communications regarding trial results for a period that does not exceed 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.